CLINICAL TRIAL: NCT05101382
Title: A Retrospective Protocol Empowering Precision Research in Colorectal Cancer (ALFAOMEGA-RETRÒ)
Acronym: ALFAOMEGA-R
Status: Recruiting | Type: Observational
Sponsor: IFOM ETS - The AIRC Institute of Molecular Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IFOM-CPO006/2019/PO005
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; CRC; Gastrointestinal disease
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE tissue Frozen biological samples (whole blood, plasma, PBMC, stools, buccal swabs, urines)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort of CRC patients: Stage-mixed cohort of at least 500 CRC patients that cannot be reached for informed consent (death or lost-to-follow-up)
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Retrospective Observation of standard clinical practice

SUMMARY:
ALFAOMEGA-RETRÒ will be exploited to retrospectively collect clinical and imaging data and archival samples to be used for validation and correlative studies on markers discovered by cutting-edge translational projects within the AIRC5x1000 program "Insights into the evolving heterogeneity of colorectal cancer (CRC): from mechanism to therapies" (an ongoing multi-institutional research program).

DETAILED DESCRIPTION:
ALFAOMEGA-RETRÒ, the retrospective "mirror" protocol of ALFAOMEGA (protocol n. IFOM-CPO003/2018/PO002), has been designed to build a retrospective collection of clinically annotated data and biological samples retrieved from colorectal cancer patients (CRC).

The repository will feed experimental precision research aimed at i) defining a new taxonomy of CRC based on evolutionary patterns (retrospectively assessed on patient's samples), ii) developing and evaluating innovative biomarker-specific therapeutic strategies derived from or together with ALFAOMEGA.

The following data and biological samples will be collected:

* Clinical Data (Demographics, Medical History, Cancer Diagnosis & History, Treatment Assessment,).
* Imaging Data (CT-Scans, MRI, PET...).
* Formalin-Fixed Paraffin-Embedded (FFPE) tissue (either from surgical resections or diagnostic biopsies).
* Frozen biological samples (blood, plasma, PBMC, stools, buccal swabs, urines, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of colorectal cancer (any stage).
* Age >18 years at the time of diagnosis.
* Availability of clinically-annotated radio-imaging data and/or diagnostic Formalin-Fixed Paraffin Embedded (FFPE) blocks (surgical resections and/or tumor biopsies), or at least 10 slides (preferably 20). FFPE tissue blocks are always preferred to slides.
* Verification that the patient could not be reached for informed consent in accordance with applicable national regulations.

Exclusion Criteria:

* if inclusion criteria are not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: at least 500 colorectal cancer patients at any stage who cannot be reached for an informed consent
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of retrospectively recruited CRC cases | 6 months
  Number of retrospectively recruited CRC cases with complete matched clinical data, radio-imaging data and FFPE or frozen biological samples.

OTHER OUTCOMES:
Number of new prognostic and predictive markers | 6 months
  Number of identified/validated new independent prognostic and predictive biomarkers
Biomarkers correlation with PFS | 6 months
  Correlation of new prognostic and predictive biomarkers with progression-free survival (PFS).
Biomarkers correlation with OS | 6 months
  Correlation of new prognostic and predictive biomarkers with overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Marsoni, MD, Study Director — IFOM ETS - The AIRC Institute of Molecular Oncology
Locations (13):
- Italy (9):
  - Ospedale Policlinico San Martino, Genova, GE
  - Fondazione IRCCS, Istituto Nazionale dei Tumori, Milan, MI
  - Niguarda Cancer Center - ASST Grande Ospedale Metropolitano Niguarda, Milan, MI
  - IRCCS Istituto Clinico Humanitas, Milan, MI
  - Istituto Oncologico Veneto (IOV), Padua, PD
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Pisa
  - Istituto di Candiolo - IRCCS, Candiolo, TO
  - Azienda Ospedaliero Universitaria San Luigi Gonzaga, Orbassano, TO
  - Azienda Ospedaliera Ordine Mauriziano, Torino, TO
- Spain (4):
  - Institut Català D'Oncologia (ICO), L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - INCLIVA - Instituto de Investigatión Sanitaria, Valencia

IPD SHARING:
Plan to Share IPD: Undecided